CLINICAL TRIAL: NCT00233363
Title: An Exploratory Study of Rebamipide to Evaluate Efficacy and Safety in the Treatment of Dry Mouth in Patients With Sjögren's Syndrome
Brief Title: Exploratory Study for Dry Mouth in Patients With Sjögren's Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 037-04-001; JapicCTI-050036
Record Dates: First submitted 2005-10-04; First posted 2005-10-05 (Estimated); Results first posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Xerostomia; Sjogren's Syndrome
MeSH Terms: conditions — Xerostomia; Sjogren's Syndrome | interventions — rebamipide

INTERVENTIONS:
Drug: Rebamipide

SUMMARY:
The purpose of this study is to exploratively investigate the clinical efficacy of rebamipide on dry mouth in patients with Sjögren's syndrome in comparison with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Sjögren's syndrome (Revised Japanese criteria for Sjögren's syndrome (1999): 1998 research report on immunological intractable diseases specified by the Japanese Ministry of Health and Welfare)
2. Patients aged 20 years or older at time of consent
3. Patients with dry mouth
4. Patients with decreased salivation

Exclusion Criteria:

1. Patients who have developed dry mouth clearly due to a cause other than Sjögren's syndrome
2. Patients in whom Saxon test cannot be performed (artificial tooth, tooth implant, etc.)
3. Patients who have received rebamipide within 3 months prior to obtaining informed consent
4. Patients who are pregnant, possibly pregnant, or lactating
5. Patients with a history of hypersensitivity to rebamipide
6. Patients who have received any other investigational drug within 3 months prior to obtaining informed consent
7. Patients who are otherwise judged inappropriate for inclusion in the study by the investigator or subinvestigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2005-04-15 (Actual); Primary Completion 2006-01-19 (Actual); Study Completion 2006-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katsuhisa Saito, Study Director — Division of New Product Evaluation and Development
Locations (1):
- Otsuka Pharmaceutical Co., Ltd., Tokyo, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Rebamipide: A rebamipide 100 mg tablet was administered orally three times a day for eight weeks.
- Placebo: A placebo tablet was administered orally three times a day for eight weeks.
Period: Overall Study
Arm/Group | Rebamipide | Placebo
Started | 53 | 51
Completed | 50 | 46
Not Completed | 3 | 5
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Aggravation of complication | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Efficacy Analysis Set comprised subjects in the Full Analysis Set (subjects received IMP at least once) excluding ineligible subjects and subjects with protocol deviations as described below:
  1. Subjects violating the rules on concomitant therapy
  2. Subjects with poor treatment compliance (<80% of the prescribed dose at time of treatment discontinuation/completion)
  3. Subjects with missing data on the primary endpoint at all time points
Groups:
- Total: Total of all reporting groups
Arm/Group | Rebamipide | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 17 | 17 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 48 | 97
  Male | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Overall Improvement Rate in Dry Mouth Symptoms
Description: At visits to the study site at two, four, and eight weeks after the start of administration, subjects self-assessed the overall change in their dry mouth symptoms in comparison with their symptoms before the start of treatment on the following four-grade scale: (1) Markedly improved (clearly better), (2) Improved (better) , (3) Unchanged (almost no difference), and (4) Aggravated (worse).
  The improvement rate was calculated by defining improvement as an assessment of either (1) Markedly improved or (2) Improved.
Time Frame: Weeks 2, 4, and 8
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rebamipide | Placebo
Number analyzed (Participants) | 50 | 50
percentage of participants
  Week 2 | 26.0 [13.8 to 38.2] | 20.0 [8.9 to 31.1]
  Week 4: number analyzed (Participants) | 50 | 48
  Week 4 | 44.0 [30.2 to 57.8] | 27.1 [14.5 to 39.7]
  Week 8: number analyzed (Participants) | 49 | 46
  Week 8 | 46.9 [33.0 to 60.9] | 39.1 [25.0 to 53.2]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from the start of IMP administration up to 9 weeks.
Description: Safety analysis set included all subjects who received investigational medicinal product (IMP) at least once and from whom data on at least 1 safety endpoint were obtained after the start of IMP administration.
Arm/Group | Rebamipide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/51
Serious Adverse Events (participants affected / at risk) | 1/53 | 1/51
Other Adverse Events (participants affected / at risk) | 31/53 | 34/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide (N=53) | Placebo (N=51)
Herpes zoster (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rebamipide (N=53) | Placebo (N=51)
Blepharitis (Eye disorders) | 0 | 1
Blepharospasm (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Conjunctivitis allergic (Eye disorders) | 0 | 1
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Oral pain (Gastrointestinal disorders) | 1 | 0
Parotid gland enlargement (Gastrointestinal disorders) | 2 | 3
Salivary gland pain (Gastrointestinal disorders) | 0 | 1
Stomach discomfort (Gastrointestinal disorders) | 0 | 1
Stomatitis (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 1 | 1
Chapped lips (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Face oedema (General disorders) | 1 | 0
Feeling abnormal (General disorders) | 1 | 1
Malaise (General disorders) | 2 | 0
Pyrexia (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Liver disorder (Hepatobiliary disorders) | 1 | 0
Furuncle (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 6
Parotitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 2
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Protein total increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 1
White blood cell count increased (Investigations) | 1 | 0
Urine bilirubin increased (Investigations) | 0 | 1
Gout (Investigations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 4
Hypoaesthesia (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 0 | 2
Intercostal neuralgia (Nervous system disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0
Pruritus genital (Reproductive system and breast disorders) | 0 | 1
Choking sensation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No